CLINICAL TRIAL: NCT07125417
Title: Non-Antithrombotic Versus. Single antiPlatelet Therapy Following Left Atrial Appendage Closure：NAPT-LAAC Randomized Controlled Trial
Brief Title: Non-antithrombotic Versus. Single Antiplatelet Therapy Following Left Atrial Appendage Closure
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: OCEAN-SHD Study Group (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAPT-LAAC trial
Record Dates: First submitted 2025-07-24; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Nonvalvular Atrial Fibrillation; Aspirin; Non-Antithrombotic Therapy; High Bleeding Risk; Left Atrial Appendage Closure
Keywords: Left Atrial Appendage Closure; High bleeding risk; Non-Antithrombotic therapy; Aspirin; Nonvalvular Artial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAPT Arm (Single Antiplatelet Therapy Arm) (Active Comparator)
  Interventions: Drug: Single Antiplatelet Therapy or No Therapy (Control)
- NAPT Arm (Non-Antithrombotic Therapy Arm) (Experimental)
  Interventions: Other: Non-Antithrombotic Therapy

INTERVENTIONS:
Drug: Single Antiplatelet Therapy or No Therapy (Control) — Monotherapy with oral anticoagulants (OAC) including direct oral anticoagulants (DOAC) and vitamin K antagonist oral anticoagulants (VKA) for 45 days after left atrial appendage closure (LAAC), followed by aspirin-directed antiplatelet monotherapy (Single Antiplatelet Therapy: SAPT) through the end of the observational period.
  Arms: SAPT Arm (Single Antiplatelet Therapy Arm)
Other: Non-Antithrombotic Therapy — Monotherapy with OAC for 45 days after LAAC, followed by no antithrombotic therapy (Non-Antithrombotic Therapy: NAPT) from enrollment through the end of the observational period.
  Arms: NAPT Arm (Non-Antithrombotic Therapy Arm)

SUMMARY:
The goal of this clinical trial is to verify that Non-Antithrombotic Therapy (NAPT) followed by Oral Anticoagulants (OAC) monotherapy for 45 days after Left Atrial Appendage Closure (LAAC) is non-inferior to Single Antiplatelet Therapy (SAPT) with aspirin during the period from randomization to the end of observational period (4 years at the maximum) in non-valvular atrial fibrillation subjects with high bleeding risk.

The primary endpoint is a composite endpoint consisting of all-cause mortality, myocardial infarction, stroke, systemic embolism, major bleeding, or clinically relevant non-fatal bleeding from randomization to the end of study observation (up to a maximum follow-up of 4 years).

* Participants will be enrolled in this study until the day following the implementation of LAAC and will be randomized to the SAPT arm and NAPT arm in a 1:1 ratio.
* Participants will be observed for 4 years from the time the first subject is enrolled in this study.
* Participants will visit the hospital at 45 days, 1 year, and 2 years after enrollment, and will also be followed up by telephone, basically at the end of the observation period (up to a maximum follow-up of 4 years).

<Study treatment duration> In both arms, OAC monotherapy will be initiated in the first 24 hours of enrollment and continued for 45 days (allowed window period: plus 2 weeks)..

* SAPT arm will continue to receive 45 days of OAC monotherapy followed by low-dose aspirin (75～100 mg/day) as an antithrombotic agent required through the end of the study observation period.
* NAPT arm do not receive antithrombotic medication after 45 days of OAC monotherapy through the end of the study observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has documented non-valvular atrial fibrillation (i.e, atrial fibrillation without severe mitral stenosis or mechanical valves)
2. Patient has CHA2DS2-VA score of 2 or greater
3. Patient meets the guidelines for proper use of the left atrial appendage closure system including patient who has an increased risk of bleeding.
4. Individual with nonvalvular atrial fibrillation who underwent successful LAAC (defined as no significant residual circumferential leak [>3 mm] or major morbidity by the time of procedure completion).
5. Patient suitable for pharmacotherapy as defined in this study protocol in both NAPT and SAPT arms
6. LAA anatomy is accommodate Boston Scientific WATCHMAN FLX Pro and LAAC procedure
7. The patient and the investigator and/or subinvestigator agree that the patient will return for all required VISITs after LAAC procedure
8. Patient has thoroughly understood the purpose of the study and has provided written informed consent to participate in the study

Exclusion Criteria:

1. Patients who are currently enrolled in other clinical trials, except when the patient is participating in a mandatory governmental registries or purely observational registries with no associated treatment.
2. Individuals require long-term anticoagulation therapy for reasons other than atrial fibrillation (AF)-related stroke risk reduction (e.g.,thrombophilic conditions, previous pulmonary embolism, or deep venous thrombosis).
3. Patients requiring oral antiplatelet therapy for reasons other than LAAC (e.g.,history of myocardial infarction, history of endovascular treatment, history of stroke/transient ischemic attack, significant coronary stenosis proven by myocardial ischemia, severe carotid stenosis requiring invasive treatment,hematologic disease such as antiphospholipid syndrome or if the investigator and/or subinvestigator judged the need for antiplatelet therapy).
4. Patients who meet one or more of the following criteria

   * Patients who are contraindicated for DOAC or VKA
   * Patients with a contraindication to aspirin
   * Patients diagnosed with an allergy to aspirin
5. Those who have or are scheduled to undergo cardiac or noncardiac intervention or surgery 45 days or 60 days before or after LAAC (e.g.,cardioversion, PCI, cardiac ablation, cataract surgery, other structural heart interventions).
6. Patients with stroke (either ischemic or hemorrhagic) or transient ischemic attack within 30 days prior to enrollment
7. Patients with active bleeding
8. Individuals who lack LAA or whose LAA has been surgically ligated
9. Individuals who experienced a myocardial infarction (with or without intervention) recorded as a non-ST elevation myocardial infarction or ST elevation myocardial infarction in the 30-day period prior to enrollment
10. Patients with previous atrial septal repair or with atrial septal defect/patent foramen ovale device
11. Patients with mechanical valve prostheses at any site
12. Persons with known contraindications to TEE
13. Patients with active infection
14. Individuals with NYHA class related IV congestive heart failure at enrollment
15. Patients who are pregnant, breastfeeding, or wishing to become pregnant
16. Patients with an expected life expectancy of less than 2 years
17. Patients requiring emergency surgery for any reason
18. Patients who, at the discretion of the investigator, have other medical, social, or psychological conditions that preclude adherence to appropriate consent or the follow-up tests required by the protocol
19. Other patients whose investigator or subinvestigator judges their participation in the study to be inappropriate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
A composite endpoint consisting of all-cause mortality, myocardial infarction, stroke, systemic embolism, major bleeding, or clinically relevant non-fatal bleeding | Through study completion, maximum of four years, with a minimum follow-up period of two years from the time of randomization.
  The definition of major bleeding or clinically significant nonfatal bleeding for the primary endpoint is BARC type 2, 3, or 5 bleeding among BARC type 1, 2, 3, 4, and 5.
  Surviving cases with no events shall be censored as of the date of discontinuation of study treatment or the date of last confirmation of survival.
  Planned enrollment term is two years, and all subjects will be obsserved until 4 years after first enrollment.

SECONDARY OUTCOMES:
Non-procedure-related BARC bleeding events of Type 1 or greater | Through study completion, maximum of four years, with a minimum follow-up period of two years from the time of randomization.
  Non-procedure-related was defined as occurring after 7 days after the LAAC procedure.
  It will be assessed throughout the entire study period, as well as from the day following Visit 1 (occurring 46 to 60 days post-randomization) until the end of the study.
ISTH major bleeding not related to the procedure and clinically relevant non-fatal bleeding | Through study completion, maximum of four years, with a minimum follow-up period of two years from the time of randomization.
  Not related to the procedure refers to events occurring 7 days after the LAAC procedure.
  It will be assessed throughout the entire study period, as well as from the day following Visit 1 (occurring 46 to 60 days post-randomization) until the end of the study.
Incidence of device-related thrombus (DRT) detected by CT and/or transesophageal echocardiography (TEE) | at Visit 1 (46~60days after randomization), 1 year, and 2 years after randomization
Combined endpoint consisting of the occurrence of ischemic stroke and systemic embolism | Through study completion, maximum of four years, with a minimum follow-up period of two years from the time of randomization.
  It will be assessed throughout the entire study period, as well as from the day following Visit 1 (occurring 46 to 60 days post-randomization) until the end of the study.

CONTACTS AND LOCATIONS:
Locations (21):
- Japan (21):
  - Nagoya Heart Center, Nagoya, Aichi-ken
  - Toyohashi Heart Center, Toyohashi, Aichi-ken
  - New Tokyo Hospital, Matsudo, Chiba
  - Kokura Kinen Hospital, Kitakyushu, Fukuoka
  - Gifu Heart Center, Gifu, Gifu
  - Medical Corporation Sapporo Heart Center Sapporo Cardio Vascular Clinic, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Tokai University Hospital, Isehara, Kanagawa
  - St.Marianna University Hospital, Kawasaki, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - The Sakakibara Heart Institute of Okayama, Okayama, Okayama-ken
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Mitsui Memorial Hospital, Chiyoda-ku, Tokyo
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - IMS Tokyo Katsushika General Hospital, Katsushika-ku, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Toyama University Hospital, Toyama, Toyama

IPD SHARING:
Plan to Share IPD: Undecided